CLINICAL TRIAL: NCT01022411
Title: A Randomized Prevention Trial Substituting Brown Rice for White Rice to Lower Markers for Diabetes Risk
Brief Title: Brown Rice Intervention on Metabolic Syndrome (BRIMS)
Acronym: BRIMS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Xu Lin, Principal Investigator, Institute for Nutritional Sciences, Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KSCX1-YW-02-BR
Record Dates: First submitted 2009-11-30; First posted 2009-12-01 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2010-10

CONDITIONS: Metabolic Syndrome X
Keywords: brown rice; white rice; diabetes risk
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Brown rice
  Interventions: Dietary Supplement: Brown rice/White rice
- B (Placebo Comparator): White rice
  Interventions: Dietary Supplement: Brown rice/White rice

INTERVENTIONS:
Dietary Supplement: Brown rice/White rice — ad libitum intake of brown rice/white rice at every lunch and dinner for 16 weeks

SUMMARY:
The specific aim of this study is to determine the effects of substituting brown for white rice on the treatment of metabolic syndrome (MetS).

DETAILED DESCRIPTION:
Metabolic syndrome (MetS), a constellation of metabolic abnormalities including central obesity, dyslipidemia, elevated blood pressure and hyperglycemia, is associated with the development of type 2 diabetes and CVD. It has become one of the major public health challenges in China due to rapidly nutrition transition and the nature of obesity epidemic. Treatment of MetS in China is very important for the prevention of the epidemic of its consequences (such as CVD and type 2 diabetes).

Compelling evidence from recent human studies has demonstrated that diet modifications are effective means in MetS management. Consumption of carbohydrate-rich foods such as rice affects blood glucose and influences diabetes risk. Specifically, eating polished white rice may increase diabetes risk, whereas eating brown rice, a whole grain product, may decrease risk. This is likely related to the different ability of white and brown rice to raise blood glucose levels, as measured by their glycemic index (GI) and glycemic load (GL), and to the higher levels of dietary fiber, vitamin B complex, magnesium and other micronutrients in brown rice.

A total of 200 participants with MetS (defined by ATP-III criteria) will be randomly assigned to a brown rice diet or an isocaloric white rice diet for 16 weeks. Effects of substituting brown for white rice will be evaluated by measuring metabolic profile (BMI, blood pressure, total cholesterol, triglyceride, LDL-C and HDL-C, fasting glucose and insulin, HbA1C).

ELIGIBILITY:
Inclusion Criteria:

* The updated National Cholesterol Education Program Adult Treatment Panel III (NCEP ATP III) criteria for the diagnosis of the MetS will be used. MetS will be defined with at least three of the following abnormalities:

  * central obesity (defined as waist circumference ≥ 80 cm for women or ≥ 90 cm for men)
  * Raised triglycerides level: ≥ 150 mg/dL (1.7 mmol/L), or specific treatment for this lipid abnormality;
  * Reduced HDL cholesterol: < 40 mg/dL (1.0 mmol/L) in males and < 50 mg/dL (1.3 mmol/L) in females, or specific treatment for this lipid abnormality;
  * Elevated blood pressure (BP): systolic BP ≥ 130 or diastolic BP ≥ 85 mm Hg, or treatment of previously diagnosed hypertension;
  * Increased fasting plasma glucose (FPG): ≥ 100 mg/dL (5.6 mmol/L), or previously diagnosed type 2 diabetes.
* Being able to comply with the specified feeding conditions
* Being able to eat brown rice
* Being between the ages of 35 and 60 years

Exclusion Criteria:

* Pregnancy or lactation
* Use of insulin
* Severe kidney disease
* Cardiovascular diseases, stroke, cancer and psychological disorders
* Brown rice allergies
* Drug or alcohol abuse

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2009-10; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
fasting glucose | 16 weeks

SECONDARY OUTCOMES:
Insulin | 16 weeks
total cholesterol | 16 weeks
triglyceride | 16 weeks
LDL-C | 16 weeks
HDL-C | 16 weeks
blood pressure | 16 weeks
HbA1c | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xu Lin, MD, PhD, Principal Investigator — Institute for Nutritional Sciecnes, Chinese Acadamy of Sciences
Locations (1):
- Institute for Nutritional Sciences, Chinese Academy of Sciences, Shanghai, China

REFERENCES:
- [Derived] Zhang G, Pan A, Zong G, Yu Z, Wu H, Chen X, Tang L, Feng Y, Zhou H, Chen X, Li H, Hong B, Malik VS, Willett WC, Spiegelman D, Hu FB, Lin X. Substituting white rice with brown rice for 16 weeks does not substantially affect metabolic risk factors in middle-aged Chinese men and women with diabetes or a high risk for diabetes. J Nutr. 2011 Sep;141(9):1685-90. doi: 10.3945/jn.111.142224. Epub 2011 Jul 27. PMID 21795429